CLINICAL TRIAL: NCT04871607
Title: A Phase 2 Trial of Yttrium-90 Labeled Anti-CD25 Monoclonal Antibody Combined With BEAM Chemotherapy (aTac-BEAM) Conditioning for Autologous Hematopoietic Cell Transplantation (AHCT) in Patients With Primary Refractory or Relapsed Hodgkin Lymphoma
Brief Title: Yttrium-90 Labeled Anti-CD25 Monoclonal Antibody Combined With BEAM Chemotherapy Conditioning for the Treatment of Primary Refractory or Relapsed Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20420; NCI-2021-03073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20420 (Other: City of Hope Medical Center); P30CA033572 (NIH); P50CA107399 (NIH)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Basiliximab; Carmustine; Cytarabine; Etoposide; pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (yttrium Y 90 basiliximab, chemotherapy, HPC-A) (Experimental): Patients receive 'cold' basiliximab IV followed by yttrium Y 90 basiliximab IV on day -14. Patients also receive carmustine IV on over 4 hours day -6, etoposide IV over 1 hours QD and cytarabine IV over 2 hours BID or QD on days -5 to -2, and melphalan IV over 1 hours on day -1. Patients then receive HPC-A product via infusion on day 0. Beginning day 5, patients receive G-CSF (or biosimilar) SC or IV until ANC > 500 for 3 consecutive days or according to the treating physician's best clinical judgement.
  Interventions: Biological: Basiliximab; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Biological: Genetically Engineered Hematopoietic Stem Progenitor Cells; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Biological: Yttrium Y 90 Basiliximab

INTERVENTIONS:
Biological: Basiliximab — Given IV
  Other Names: SDZ-CHI-621; Simulect
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Biological: Genetically Engineered Hematopoietic Stem Progenitor Cells — Given via infusion
  Other Names: Genetically Engineered HSPCs
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given SC or IV
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF
Biological: Yttrium Y 90 Basiliximab — Given IV
  Other Names: 90Y Basiliximab; Yttrium Y 90-DOTA-Basiliximab

SUMMARY:
This phase II trials studies the effects of yttrium-90 labeled anti-CD25 monoclonal antibody combined with BEAM chemotherapy conditioning in treating patients with Hodgkin lymphoma that does not response to treatment (refractory) or has come back (relapsed). Yttrium-90-labeled anti-CD25 is an antibody (proteins made by the immune system to fight infections) that is attached to a radioactive substance and may kill cancer cells and shrink tumors. Chemotherapy drugs, such as carmustine, etoposide, cytarabine, and melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a peripheral blood stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the anti-lymphoma activity of the aTac-carmustine (BCNU), etoposide, cytarabine (cytosine arabinoside), and melphalan (BEAM) regimen as conditioning for autologous hematopoietic cell transplantation (AHCT); assessed by 2-year progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. Estimate the overall survival (OS) probability and cumulative incidence of relapse/progression, and non-relapse mortality (NRM) at 100-days, 1-year and 2-years.

II. Summarize toxicities by type, frequency, severity, attribution, time course and duration.

III. Evaluate short and long-term complications, including: delayed engraftment (neutrophil and platelet), infection, and myelodysplasia (MDS).

EXPLORATORY OBJECTIVES:

I. Evaluate potential changes in Hodgkin lymphoma biological markers of patients treated with 90Y basiliximab BEAM via analyses of serial blood samples.

II. Assess the potential association between pre-AHCT CD25 expression levels and post-AHCT outcomes.

OUTLINE:

Patients receive 'cold' basiliximab intravenously (IV) followed by yttrium Y 90 basiliximab IV on day -14. Patients also receive carmustine IV on over 4 hours day -6, etoposide IV over 1 hours once daily (QD) and cytarabine IV over 2 hours twice daily (BID) or QD on days -5 to -2, and melphalan IV over 1 hours on day -1. Patients then receive hematopoietic progenitor cell apheresis (HPC-A) product via infusion on day 0. Beginning day 5, patients receive granulocyte colony-stimulating factor (G-CSF) (or biosimilar) subcutaneously (SC) or IV until absolute neutrophil count (ANC) > 500 for 3 consecutive days or according to the treating physician's best clinical judgement.

After completion of study treatment, patients are followed up at 30 days, up to 2 years for response, and up to 5 years for survival.

ELIGIBILITY:
Inclusion Criteria Informed Consent and Willingness to Participate 1. Documented informed consent of the participant and/or legally authorized representative.

- Assent, when appropriate, will be obtained per institutional guidelines Age Criteria, Performance status

1. Age: ≥18 years
2. Karnofsky performance status ≥ 70%
3. Life expectancy ≥ 6 months Nature of Illness and Illness Related Criteria
4. Histologically confirmed HL
5. High risk relapsed or refractory HL disease defined as having any one of the following:

   * B symptoms at relapse
   * Extranodal disease at relapse
   * Primary refractory disease'
   * Relapse < 1 year after completion of frontline therapy
   * Not in CR at the time of transplant
   * Relapse after receiving PD1 blockade or brentuximab vedotin as initial therapy
6. Patients will be enrolled after collection of at least 2.0 x 106 CD34 cells/kg of autologous hematopoietic progenitor cells (HPC-A) by apheresis.
7. Recovery from non-hematologic toxicities of salvage cytoreductive chemotherapy to ≤ grade 2 (CTCAE v5).

   Clinical Laboratory and Organ Function Criteria (To be performed prior to Day 1 of protocol therapy)
8. Serum creatinine ≤ 1.5 mg/dL
9. Creatinine clearance of ≥ 60 mL/min per 24 hour urine test
10. Total bilirubin ≤ 1.5 X ULN (unless has Gilbert's disease)
11. AST/SGOT ≤1.5 x ULN (except in cases where abnormal LFTs are due to involvement with HL)
12. ALT/SGPT ≤ 1.5 x ULN (except in cases where abnormal LFTs are due to involvement with HL)
13. Left ventricular ejection fraction (LVEF) ≥ 50%
14. FEV1 > 65% of predicted measured, or DLCO (diffusion capacity) ≥ 50% of predicted measured (corrected for hemoglobin).

    Contraception
15. Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least six months after the last dose of protocol therapy.

    * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria Prior and concomitant therapies

1. Planned BV consolidation after AHCT
2. Prior high dose chemotherapy with autologous stem cell transplant, or prior allogeneic transplantation.
3. Significant prior external beam dose-limiting radiation to a critical organ based on review of the prior radiation treatment records by the Radiation Oncology PI.
4. Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy.

   Other illnesses or conditions
5. Myelodysplasia or any active malignancy other than HL, or < 5 years remission from any other prior malignancy, except non-melanoma skin cancer, localized prostate cancer or localized cervical cancer
6. Any cytogenetic abnormality in the bone marrow that is known to be associated with or predictive of myelodysplasia is excluded. This includes, but is not limited to, del(5), del(7), del(11).
7. Lymphocyte-predominant Hodgkin Lymphoma
8. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 90Y-basiliximab-DOTA.
9. Persistent marrow involvement (>10%) with HL after salvage cytoreductive therapy and before stem cell mobilization.
10. BM harvest required to reach adequate cell dose for transplant.
11. Active Hepatitis B or C viral infection or Hepatitis B surface antigen positive
12. Positive Human Immunodeficiency Virus antibody, patients with undetectable HIV viral load with CD4 ≥ 300 and are on HAART medication are allowed
13. Patients should not have any uncontrolled illness including ongoing or active infection.
14. Patients with psychosocial circumstances or illnesses that preclude protocol participation (to be determined by P.I.)
15. Pregnant women are excluded from this study because 90Y-basiliximab/DOTA is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother 90Y-basiliximab/DOTA, breastfeeding should be discontinued if the mother is treated with 90Y-basiliximab/DOTA.
16. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.

    Noncompliance
17. Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

    * Eligibility should be confirmed per institutional policies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2029-10-02 (Estimated); Study Completion 2029-10-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From the start of treatment up to 5 years post transplant
  Disease relapse or progression, or death from any cause, whichever occurs first.
  Will be calculated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall survival | From the start of treatment up to 5 years post transplant
  Death from any cause. Will be calculated using the Kaplan-Meier method.
Relapse or progression | From the start of treatment up to 5 years post transplant
  Relapse or progression of Hodgkin lymphoma.
Non-relapse mortality | From the start of treatment up to 5 years post transplant
  Death from causes other than relapse or progression.
Incidence of toxicities and adverse events | Day -14 to day 100 post-transplant
  Toxicity information recorded will include the type, severity, and the probable association with the study regimen. Tables will be constructed to summarize the observed incidence by severity and type of toxicity. Toxicities will be recorded using both the Bearman criteria and the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 scale.
Time to hematopoietic recovery | Up to day 100 post transplant
  Time to neutrophil recovery will be the first of three consecutive days of ≥ 500 neutrophils/μL following the expected nadir. Time to platelet engraftment will be the first day of the first of three consecutive daily laboratory values when the platelet count is ≥20,000/μL, without a platelet transfusion in the previous seven days.
Incidence of infection | Day -14 to day 100 post-transplant
  Microbiologically documented infections will be reported by site of disease, date of onset, severity and resolution, if any.
Rate of secondary myelodysplastic syndrome | From the start of treatment up to 5 years post transplant
  Secondary MDS or AML post therapy

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States